CLINICAL TRIAL: NCT00606164
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Groups, Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Bryostatin 1 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics Study of Bryostatin 1 in Patients With Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blanchette Rockefeller Neurosciences Insitute (Other)
Responsible Party: Mark A. Cochran, Ph.D./CEO and Executive Director, Blanchette Rockefeller Neurosciences Insitute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRY-201
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; bryostatin 1; bryostatin; safety; efficacy; pharmacokinetics; pharmacodynamics; protein kinase C
MeSH Terms: conditions — Alzheimer Disease | interventions — Bryostatins; Injections; bryostatin 1; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 10 ug/m2 Bryostatin (Experimental)
  Interventions: Drug: Bryostatin for Injection
- 15 ug/m2 Bryostatin (Experimental)
  Interventions: Drug: Bryostatin for Injection

INTERVENTIONS:
Drug: Bryostatin for Injection — A single one-hour intravenous infusion of 10 or 15 ug/m2 Bryostatin for Injection on Day 1
  Other Names: Bryostatin 1; Bryostatin; NSC 339555; CAS No. 83314-01-6
  Arms: 10 ug/m2 Bryostatin; 15 ug/m2 Bryostatin
Drug: Placebo — A single one-hour intravenous infusion of placebo on Day 1
  Other Names: PET (60/30/10) diluent plus sodium chloride for injection
  Arms: Placebo

SUMMARY:
The main purpose of this study is find out how safe a single dose of bryostatin 1 is in patients with Alzheimer's Disease (AD). This study is also being done 1) to determine how effective a single dose of bryostatin 1 is in the treatment of AD, 2) to find out what happens to bryostatin 1 once it enters the body by measuring the levels of bryostatin 1 in blood, and 3) to measure a substance in the blood (protein kinase C) that may help to better understand how bryostatin 1 works.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 50 yrs or older. Females must be of non-childbearing potential (surgically sterilized or at least 2 yrs post-menopausal)
* Must have a cognitive deficit present for at least 1 yr & meet DSM-IV-TRTM criteria for AD & meet NINCDS/ADRDA criteria for the presence of probable AD
* Severity of AD must be mild to moderate, documented with a MMSE score of 12-26
* Has a CT scan or MRI scan within the prior 12 months, which is compatible with a diagnosis of probable AD
* Ability to walk, at least with an assistive device
* Vision & hearing sufficient to comply with testing
* Normal cognitive & social functioning prior to onset of dementia
* Consistent caregiver to accompany patient to assessment visits
* Sufficient basic education to be able to complete the cognitive assessments
* Living outside an institution
* Informed consent signed & dated by patient or legal representative
* Has provided written authorization for the use & disclosure of protected health information

Exclusion Criteria:

* Dementia due to any condition other than AD, including vascular dementia (modified Hachinski Ischemic Scale ≥ 5; positive NINDS-AIREN criteria)
* Evidence of clinically significant unstable cardiovascular, renal, hepatic, gastrointestinal, neurological, or metabolic disease within the past 6 months (as determined by medical history, ECG results, chest x-ray, or physical examination)
* Use of any drug within 14 days prior to randomization unless the dose of the drug & the condition being treated have been stable for at least 30 days & are expected to remain stable during the study & neither the drug nor the condition being treated is expected to interfere with the study endpoints
* Any medical or psychiatric condition that may require medication or surgical treatment during the study
* Life expectancy less than 6 months
* Any other screening laboratory values outside the normal ranges that are deemed clinically significant by the investigator
* Use of an investigational drug within 30 days prior to the screening visit or during the entire study
* Significant neurological disease other than AD, including cerebral tumor, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, & other entities
* Major depression according to DSM-IV
* Psychotic episodes requiring hospitalization or antipsychotic therapy for more than 2 weeks within the past 10 yrs, not linked to AD
* Agitation sufficient to preclude participation in this trial
* Alcohol or drug dependence diagnosed within the past 10 yrs
* Epilepsy or anti-epileptic drug therapy
* Abnormal laboratory tests that might point to another etiology for dementia: serum B12, folate, thyroid functions, electrolytes, syphilis serology
* Musculoskeletal diseases that could interfere with assessment
* Acute or poorly controlled medical illness: blood pressure> 180 mmHg systolic or 100 mmHg diastolic; myocardial infarction within 6 months; uncompensated congestive heart failure (NYHA Class III or IV), severe renal, hepatic or gastrointestinal disease that could alter drug pharmacokinetics; blood glucose > 180 mg/dl on repeated testing at entry into study or need for insulin therapy
* Previous randomization in this trial or participation in another investigational trial < 2 months prior to randomization
* Likelihood, according to clinical judgment, of being transferred to a nursing home within 6 months
* Change in dosage of any concomitant antidepressant within 30 days prior to randomization
* Lack of caregiver
* Pregnant or lactating females
* Patients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedures outlined in this protocol
* HIV positive
* Hepatitis B or C positive
* Concomitant use of medications other than AD or antidepressant medications for which the dose regimens are stabilized for at least 30 days prior to enrollment in study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 4-weeks
Alzheimer's Disease Assessment Scale | 4-weeks post dose
Clinician's Interview Based Impression of Change | 4-weeks post dose

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale | 24, 48, and 72 hrs post dose
Clinician's Interview Based Impression of Change | 24, 48, and 72 hrs post dose
Clinical Dementia Rating Battery | 24, 48, and 72 hrs post dose and 4-weeks post dose
Alzheimer's Disease Cooperative Study - Activities of Daily Living | 24, 48, and 72 hrs post dose and 4-weeks post dose
Severe Impairment Battery | 24, 48, and 72 hrs post dose and 4-weeks post dose
Hopkins Verbal Learning Test-Revised | 24, 48, and 72 hrs post dose and 4-weeks post dose
Temperature | 48 hrs and 4-weeks post dose
Respiratory rate | 48 hrs and 4-weeks post dose
Blood pressure | 15, 30, and 60 minutes after start of study drug infusion, and at 1, 2, 4, 8, 12, 24, 48, and 72 hrs post infusion and 4-weeks post infusion
Heart rate | 15, 30, and 60 minutes after start of study drug infusion, and at 1, 2, 4, 8, 12, 24, 48, and 72 hrs post infusion and 4-weeks post infusion
Electrocardiogram | 15, 30, and 60 minutes after start of study drug infusion, and at 1, 2, 4, 8, 12, and 24 hrs post infusion and 4-weeks post infusion
Physical Exam | 48 hrs and 4-weeks post dose
Hematology | 48 hrs and 4-weeks post dose
Blood chemistry | 48 hrs and 4-weeks post dose
Urinalysis | 48 hrs and 4-weeks post dose
Pharmacokinetics | Blood draws at baseline, during the study drug infusion (15, 30, and 60 minutes after start of infusion), and at 20 minutes, 1 hr, 2 hrs, 6 hrs, 24 hrs, 48 hrs, and 72 hrs post infusion
Protein kinase C activity (pharmacodynamics) | Blood draws at baseline, during the study drug infusion (15, 30, and 60 minutes after start of infusion), and at 20 minutes, 1 hr, 2 hrs, 6 hrs, 24 hrs, 48 hrs, and 72 hrs post infusion

CONTACTS AND LOCATIONS:
Overall Officials: James M Stevenson, MD, Principal Investigator — West Virginia University Department of Behavioral Medicine and Psychiatry
Locations (1):
- Chestnut Ridge Center West Virginia University Department of Behavioral Medicine and Psychiatry, Morgantown, West Virginia, United States